CLINICAL TRIAL: NCT00353145
Title: A Phase II Study to Evaluate the Efficacy and Toxicity of Oxaliplatin in Combination With Gemcitabine as First and Second Line Therapy in Unknown Primary Cancer
Brief Title: Gemox as First and Second Line Therapy in Unknown Primary Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0946
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Unknown Primary Neoplasms
Keywords: Unknown Primary Neoplasms; UPC; Unknown Primary Cancer; Questionnaire; Gemcitabine; Gemcitabine Hydrochloride; Gemzar; Oxaliplatin; Eloxatin; Gemox
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Gemcitabine; Oxaliplatin; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + Oxaliplatin (Experimental): Gemcitabine 1000 mg/m^2, infused at 10 mg/m^2/min on Day 1 and Oxaliplatin 100 mg/m^2 by vein infused on Day 2 over two hours. Repeated every 14 days (one cycle).
  Interventions: Drug: Gemcitabine (Gemox); Drug: Oxaliplatin; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Gemcitabine (Gemox) — 1000 mg/m^2, infused at 10 mg/m^2/min on Day 1 repeated every 14 days (one cycle).
  Other Names: Gemcitabine Hydrochloride; Gemzar
Drug: Oxaliplatin — 100 mg/m^2 by vein infused on Day 2 over two hours, repeated every 14 days (one cycle).
  Other Names: Eloxatin
Behavioral: Questionnaire — Quality of Life Surveys

SUMMARY:
Primary objectives:

1. To determine the overall tumor response rate with oxaliplatin in combination with gemcitabine (GEMOX) as first line and second line therapy in unknown primary cancer (UPC).
2. To determine the tolerability (toxicity) of this regimen in this patient population.

Secondary objectives:

1. To determine the median overall survival (OS) and time to progression (TTP) for patients treated with this combination.
2. To determine the impact of this combination on quality of life (QOL) in this patient population.

DETAILED DESCRIPTION:
Oxaliplatin is a chemotherapy drug that causes the death of cancer cells and other actively dividing cells by interfering with Deoxyribonucleic acid (DNA) function. Gemcitabine prevents cells from making DNA and Ribonucleic acid (RNA) that are necessary for cell growth, thus disrupting the growth of the cancer cells, which causes the cancer cells to start to die.

After the screening portion of the study, if you are eligible to begin study treatment, you will come to M. D. Anderson at least every two weeks (14 days) for treatment. Each 14-day period of treatment is called a "cycle" of therapy. You will receive at least 3 cycles of therapy (6 weeks) unless side effects become intolerable or the disease progresses.

When you begin treatment, you will have a small tube (central venous line) inserted into a large vein under the skin of the chest or through a vein in the arm for administration of oxaliplatin and gemcitabine. The central venous line will remain in place the entire time you are taking part in this study. Both drugs must be given at M. D. Anderson. On Day 1 of each cycle, you will receive gemcitabine injected into a vein over 2 hours. On Day 2 of each cycle you will receive oxaliplatin injected into a vein over 2 hours. This drug schedule will be repeated every 2 weeks.

You will first be asked to fill out several questionnaires that deal with your quality of life. These will help the researchers understand how the study drugs affect your quality of life including your pain level, fatigue (tiredness) level, appetite, and ability to perform everyday tasks, in spite of whether there is any shrinkage of the tumor. It will take about 30 minutes to an hour to complete the forms. You will also be asked to complete a questionnaire (one time only) that asks questions about why you decided to take part in this study.

During the first cycle of therapy, blood (about 2 1/2 teaspoons) will be collected once a week for routine tests. Before each new cycle of therapy, you will have a complete physical exam, urine will be collected, and blood will be drawn (about 2 ½ teaspoons) for routine tests. You will be asked to tell the study doctor about all medications you have taken since you started taking the study drugs and any health problems that you may have experienced. You will also have either computed tomography (CT) scans or an Magnetic resonance imaging (MRI) of the tumor(s) every 6 weeks and at the end of the study.

All tests before each new cycle of treatment and when treatment stops must be done at M. D. Anderson. Extra tests may be done during the study if your doctor feels it is necessary for your care. Every 6 weeks for as long as you are on study, you will also be asked to fill out the questionnaires that help study doctors understand your quality of life. It will take about 30 minutes to an hour to complete the forms.

If you experience intolerable side effects, treatment may be delayed, stopped, or you may receive smaller doses of the treatment. You may continue to receive treatment on this study, unless the disease gets worse or you experience any intolerable side effects. If this happens, you will be taken off the study and your doctor will discuss other treatment options with you.

When you stop taking part in the study for any reason, you will have blood (about 3 teaspoons) collected for final routine tests. You will have one more physical exam and either a CT scan or a MRI to check on the status of the disease. You will also be asked once more to fill out the questionnaires that help assess your quality of life. It will take about 30 minutes to an hour to complete the forms.

Once you stop receiving study treatment, you will be contacted by phone every three months for the rest of your life to check on how you are doing and any symptoms you may be experiencing.

This is an investigational study. Oxaliplatin is FDA approved for treatment of advanced cancer of the colon or rectum, and gemcitabine is FDA approved for the treatment of advanced cancer of the pancreas. However, the combination of the two drugs for treatment of cancers with unknown primaries is still considered investigational. Up to 81 people will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years old.
2. Signed informed consent/authorization is obtained prior to conducting any study-specific screening procedures.
3. Patients should fulfill the criteria for UPC: no primary detected after a complete evaluation which is defined as complete history and physical, detailed laboratory examination, directed radiologic studies, symptom or sign directed invasive studies, directed immunohistochemistry studies and serum tumor markers.
4. Previously untreated or has received no more than one prior chemotherapy regimen for unknown primary cancer. If the patients are previously treated, they may not have had previous exposure to gemcitabine or oxaliplatin. Prior exposure to cisplatin or carboplatin is allowed for this study.
5. ECOG performance status must be 0-2 (Appendix A).
6. Adequate hepatic, renal and bone marrow function: Leukocytes >= 3,000/uL; Absolute neutrophil count >= 1,500/uL; Platelets >= 100,000/uL; Total bilirubin <= 1.5 * institutional upper limits of normal (ULN); AST (SGOT)/ALT (SGPT) <= 2.5 * institutional ULN; Creatinine <= 1.5 mg/dL.
7. Women of childbearing potential are not excluded from this study; however all participants (men and women) with reproductive potential must practice an effective method of contraception while on this study in order to minimize risks to fetuses.
8. Patients may have received prior radiation treatment but the last fraction of radiation treatment must have been completed at least 4 weeks prior to entry on this study.
9. Patients must have at least one measurable lesion as per the RECIST Criteria that can be accurately measured in at least one dimension, with minimum lesion size equal to or more than twice the thickness of the imaging study used. If radiation was previously received, measurable disease must occur outside the previous radiation field, unless disease progression has been documented.
10. Both men and women and members of all ethnic groups are eligible for this trial.

Exclusion Criteria:

1. In previously treated patients; patients should not have received gemcitabine or oxaliplatin as one of the agents.
2. Uncontrolled intercurrent illness including, but not limited to, active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmias not well controlled with medication, myocardial infarction within the previous 6 months, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events. A CT scan of the brain is not needed for eligibility and will be done only if the patient presents with symptoms suggestive of brain metastases.
4. Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 28 days earlier.
5. Patients may not be receiving any other investigational agents, or have participated in any investigational drug study within 28 days preceding start of study treatment.
6. The teratogenic potential of this combination is currently unknown. Women who are pregnant or lactating are excluded.
7. History of any other malignancy in the last 5 years, except patients with a prior history of in situ cancer or basal or squamous cell skin cancer are eligible.
8. Peripheral neuropathy > grade 1.
9. Female patients with adenocarcinoma with axillary only nodes will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-02; Primary Completion 2007-03 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Participants' Response | Response to treatment measured using Response Evaluation Criteria in Solid Tumors (RECIST) criteria with radiological evaluation at 6 weeks and reevaluated every 6 weeks.
  Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least 30% decrease in sum of longest diameter (LD) of target lesions, reference baseline sum LD; Progressive Disease (PD): At least 20% increase in sum of LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of 1 or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor increase to qualify for PD, reference smallest sum LD since treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: Gauri R. Varadhachary, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Carlson H, Lenzi R, Raber MN, Varadhachary GR. A phase II study to evaluate the efficacy and toxicity of oxaliplatin in combination with gemcitabine in carcinoma of unknown primary. Int J Clin Oncol. 2013 Apr;18(2):226-31. doi: 10.1007/s10147-011-0366-4. Epub 2012 Jan 5. PMID 22218909
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org